CLINICAL TRIAL: NCT03292224
Title: Systemic Fungal Infections in Intensive Care Unit Patients
Brief Title: Systemic Fungal Infections in ICU Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Selim, Resident Doctor, Assiut University
Other Study IDs: SFI in ICU Patients
Record Dates: First submitted 2017-08-29; First posted 2017-09-25 (Actual); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Microscopy; Diagnostic Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: - Microscopic examination and culture of collected specimens — 1. Unstained wet mount with 10%-20% KOH.
  2. Wet mounts stained with:
     * Lactophenol cotton blue.
     * India ink
     * Gram stain Culturing on Sabouraud´s dextrose agar .
  Other Names: • Complete blood picture and Chest radiography.

SUMMARY:
This study aims to :

1. Diagnosis of Systemic fungal infections in ICU patients.
2. Detection the most common fungal species in ICU.
3. Detection of in vitro antifungal sensitivity pattern

DETAILED DESCRIPTION:
Systemic fungal infections are a significant and growing public health problem ,Over the past few years, major advances in healthcare have led to an unwelcome increase in the number of life-threatening infections due to true pathogenic and opportunistic fungi ,These have a significant impact on morbidity, mortality, length of hospital stay, and healthcare costs in critically ill patients in intensive care unit ( ICU).

Health care workers encounter at risk patients in ICU in various settings : including diabetes mellitus, renal insufficiency, surgery (especially abdominal surgery), the use of broad-spectrum antibiotics, parenteral nutrition, hemodialysis, mechanical ventilation, the presence of central vascular catheters, and therapy with immunosuppressive agents,Prolonged treatment with corticosteroids before ICU admission, liver cirrhosis with prolonged ICU stay (.7 days), solid organ cancer, HIV infection and lung transplantation are also considered as risk factors ,It can also occur following trauma or invasion of wounds covered with contaminated dressings, e.g. in the ICU. One outbreak of gastric mucormycosis in ICU patients reported in Spain arose in association with the use of contaminated wooden tongue depressors in critically ill patients.

Candida and Aspergillus species are the most frequent causes of healthcare-associated fungal infections in these patients, Although Candida infections are the most frequent fungal infections in ICU patients, invasive aspergillosis is associated with higher morbidity and mortality rates even in the absence of traditional risk factors,Invasive candidiasis is a highly lethal infection associated with mortality rates between 40 and 60 %. The five most common Candida species are Candida albicans, Candida glabrata, Candida tropicalis, Candida parapsilosis, and Candida krusei.

Accurate diagnosis of invasive fungal infection is crucial so that appropriate antifungal agents can be started rapidly. However, early diagnosis is not always easy. Microscopic examination is rapid and can be helpful but a negative result does not exclude infection. Blood cultures are positive in only 50-70 % of cases of Candida BSI, Furthermore, it can take several days before Candida is identified at the species level and antifungal susceptibility data are available but remain the gold stander in diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Suppressed immunity such as: (patients with malignancy under chemotherapy, prolonged use of corticosteroids.………etc)
* Manifestations of chest infection e.g.cough, Haemoptysis, dyspnea and chest discomfort.
* Persistent fever resistant to antibiotic therapy.
* Urinary manifestations resistant to antibiotic therapy.

Exclusion Criteria:

* Patients who received antifungal therapy within 3 days prior to sample collection.
* Patients refused to participate in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will include patients who will be admitted to intensive care unit in Assiut University Hospital regardless to age and sex.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09-28 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-10-15 (Estimated)

PRIMARY OUTCOMES:
Positive cultures of collected specimens from patients in ICU with suspected SFI. | 2weeks
  samples (blood ,urine and sputum) will be taken under complete aseptic precautions in sterile containers and carried immediately for culturing on sabouraud dextrose agar .Positive cultures help in early diagnosis of systemic fungal infections

REFERENCES:
- [Background] Jensen J, Guinea J, Torres-Narbona M, Munoz P, Pelaez T, Bouza E. Post-surgical invasive aspergillosis: an uncommon and under-appreciated entity. J Infect. 2010 Feb;60(2):162-7. doi: 10.1016/j.jinf.2009.11.005. Epub 2009 Nov 20. PMID 19932132
- [Background] Leleu G, Aegerter P, Guidet B; College des Utilisateurs de Base de Donnees en Reanimation. Systemic candidiasis in intensive care units: a multicenter, matched-cohort study. J Crit Care. 2002 Sep;17(3):168-75. doi: 10.1053/jcrc.2002.35815. PMID 12297992
- [Background] Pappas PG, Kauffman CA, Andes DR, Clancy CJ, Marr KA, Ostrosky-Zeichner L, Reboli AC, Schuster MG, Vazquez JA, Walsh TJ, Zaoutis TE, Sobel JD. Clinical Practice Guideline for the Management of Candidiasis: 2016 Update by the Infectious Diseases Society of America. Clin Infect Dis. 2016 Feb 15;62(4):e1-50. doi: 10.1093/cid/civ933. Epub 2015 Dec 16. PMID 26679628
- [Background] O'Keefe SJ, Sender PM, Clark CG, James WP. Proceedings: The dynamics of protein metabolism following operative trauma. Clin Sci Mol Med. 1974 Sep;47(3):15P. doi: 10.1042/cs047015pa. No abstract available. PMID 4419464